CLINICAL TRIAL: NCT06669182
Title: Effects of Cerebellar Transcranial Magnetic Stimulation on Patients With Alzheimer's Disease：A Multicenter Randomized Controlled Trial
Brief Title: Advantage of Cerebellar Transcranial Magnetic Stimulation in Alzheimer's Diseases （ACT-AD）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20242285jiangwen
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease; Transcranial Magnetic Stimulation; Cerebellum
Keywords: Transcranial magnetic stimulation; Intermittent theta burst stimulation; Cerebellar cognitive reserve; Default mode network; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (Active Comparator): Participants will receive iTBS-TMS once a day for 4 weeks, followed by once a week for 8 weeks.
  Interventions: Device: Intermittent Theta-Burst Transcranial Magnetic Stimulation
- Assigned Interventions (Sham Comparator): Participants will receive sham iTBS-TMS once a day for 4 weeks, followed by once a week for 8 weeks.
  Interventions: Device: Intermittent Theta-Burst Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Intermittent Theta-Burst Transcranial Magnetic Stimulation — 50Hz, stimulation intensity of 100% RMT, duration of 40s as a group of stimulation, 600 stimulation pulses, repeated stimulation of bilateral cerebellar dentate nuclei, with a 5-minute interval between each group, 1200 stimulation pulses per site, 5 times a week, treatment for 4 weeks, then treat once a week for 8 weeks.

SUMMARY:
Alzheimer's Disease (AD) is the primary cause of dementia, with its prominent feature being cognitive decline. The cerebellum plays a crucial role in cognitive processing, making it a potential target for therapeutic intervention. This study will be conducted to evaluate the efficacy and safety of cerebellar Intermittent theta-burst stimulation (CRB-iTBS) in participants with mild Alzheimer's disease on the change from baseline in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) at 3 months of treatment in the Core Study. This project aims to provide a valid treatment to improve the cognitive function and quality of life for those with Alzheimer's disease.

DETAILED DESCRIPTION:
Background:

Alzheimer's disease (AD) is a progressive neurodegenerative disease that poses substantial challenges for both families and society. The primary pathological hallmarks of AD are β-amyloid plaque (Aβ) deposition and neurofibrillary tangles. Notably, the cerebellum seems to be resilient to these pathological developments in the initial phases of AD. This early resistance of the cerebellum suggests it might contribute to compensating for the cognitive impairments associated with AD. Enhancing cerebellar reserve is a potential therapeutic approach. Repetitive transcranial magnetic stimulation (rTMS) has been explored as a means to achieve this, attributed to synaptic plasticity in the cerebellar cortex.

Hypothesis:

The cerebellar dentate nucleus (CDN), a crucial node for information transmission between the cerebellum and cerebral cortex, shows abnormal functional connectivity with cortex in AD patients. Preclinical studies demonstrated that stimulating lateral cerebellar nucleus, the rodent homologue of the human CDN, enhanced cognitive rehabilitation and improved cortical plasticity in animals after brain injury, suggesting CDN as a neuromodulation target for cognitive networks. We speculate that intermittent θ-burst stimulation (iTBS) based TMS targeting the cerebellar dentate nucleus may improve cognitive function, brain function, and lymphatic drainage in AD patients.

Specific aims:

In this study, we will conduct a randomized, double-blind, sham-controlled clinical trial focusing on the cerebellum with iTBS to assess its efficacy, safety and potential mechanisms in the treatment of AD patients. The findings yielded by the present project will have a potential strong impact on clinical practice of AD patients. Since rTMS is well tolerated and relatively low-priced, a positive result could lead to a fast application of the present proposal to the clinical experience. If successful, the proposed project will provide support for a novel treatment for cognitive dysfunction in AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50-85 years old
2. Meet the core clinical criteria of NIA-AA for possible Alzheimer's disease dementia, and PET or cerebrospinal fluid markers show elevated p-tau and decreased A β (1-42)
3. MMSE score ranges from 18-26 points; CDR score 0.5-1 points
4. The patient has received treatment with acetylcholinesterase inhibitors (AChEI), NMDA receptor antagonists, or mannequine therapy, and the current dosing regimen has remained stable for the 12 weeks prior to baseline assessment
5. At least one adult caregiver
6. The patient or legal guardian voluntarily signs the informed consent form

Exclusion Criteria:

1. Neurodegenerative disorders other than AD.
2. Significant intracranial focal or vascular pathology seen on brain MRI scan
3. History of seizure (with the exception of febrile seizures in childhood)
4. Any of the following psychotic disorders (DSM IV-TR criteria):

   * Major depressive disorder (current)
   * Schizophrenia
   * Other psychotic disorders, bipolar disorder, or substance related disorders (within the past 5 years)
5. GDS score ≥ 8 points in baseline assessment
6. Cerebrovascular disease, severe infection, malignant tumor, or severe dysfunction of organs such as heart, liver, and kidney.
7. Pregnant or lactating women
8. Contraindications for TMS or MRI, metal or implanted devices in the body (such as pacemakers, deep brain stimulators).
9. Participate in AD related clinical trials within 6 months prior to research registration

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
The changes in CDR-SB（Clinical Dementia Rating-Sum of Boxes） | baseline, 12 weeks after start of the treatment
  The changes in CDR-SB will constitute the major research outcome measure used to assess response to rTMS.There are two scoring methods for the CDR scale, namely Total Score Calculation (CDR-GS) and Sum of Six Content Calculation (CDR-SB). The scoring method used in this study is CDR-SB, with a total score of 18 points. The lower the score, the milder the symptoms

SECONDARY OUTCOMES:
The changes in MMSE（Mini Mental State Examination） | baseline, 12 weeks ,24 weeks and 36 weeks after start of the treatment
  The changes in MMSE will constitute the secondary research outcome.The full name of MMSE is mini-mental state examination. The higher the score, the better. In this study, changes in MMSE scores before and after treatment were used as secondary observations.
The changes in ADCS-ADL（Alzheimer's Disease Cooperative Study - Activities of Daily Living） | baseline, 12 weeks, 24 weeks and 36 weeks after start of the treatment
  ADCS-ADL total score is 54 points, the higher the score，the lighter the symptoms.
The changes in NPI（Neuropsychiatric Inventory） | baseline, 12 weeks, 24 weeks and 36 weeks after treatment
  The changes in NPI will constitute the secondary research outcome. The Neuropsychology Scale (NPI) evaluates 12 neuropsychiatric disorders which included 10 neuropsychiatric symptoms and 2 autonomic neurological symptoms based on the caregiver's perception of the patient's behavior and the perceived distress. The lower the score, the lighter the symptoms.
The changes in MRI（Magnetic Resonance Imaging） | baseline and 12 weeks after treatment
  This study mainly applied resting blood oxygen level dependent functional magnetic resonance imaging (BOLD), arterial spin labeling (ASL), and magnetic resonance diffusion tensor imaging (DTI) techniques to evaluate the changes in functional connectivity of the cerebellar dentate nucleus in healthy subjects and patients before and after 12 weeks of TMS treatment, as well as the changes in the cerebellar cortical white matter fiber bundles two month after treatment.
The changes in CDR-SB（Clinical Dementia Rating-Sum of Boxes） | 24 weeks and 36 weeks after start of the treatment
  The changes in CDR-SB will constitute the major research outcome measure used to assess response to rTMS.There are two scoring methods for the CDR scale, namely Total Score Calculation (CDR-GS) and Sum of Six Content Calculation (CDR-SB). The scoring method used in this study is CDR-SB, with a total score of 18 points. The lower the score, the milder the symptoms

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Tangdu Hospital of Air Force Military Medical University, Xi'an, Shannxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shannxi
  - The Third Hospital of Xi'an, Xi'an, Shannxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooperrider J, Furmaga H, Plow E, Park HJ, Chen Z, Kidd G, Baker KB, Gale JT, Machado AG. Chronic deep cerebellar stimulation promotes long-term potentiation, microstructural plasticity, and reorganization of perilesional cortical representation in a rodent model. J Neurosci. 2014 Jul 2;34(27):9040-50. doi: 10.1523/JNEUROSCI.0953-14.2014. PMID 24990924
- [Result] Pezzetta R, Gambarota F, Tarantino V, Devita M, Cattaneo Z, Arcara G, Mapelli D, Masina F. A meta-analysis of non-invasive brain stimulation (NIBS) effects on cerebellar-associated cognitive processes. Neurosci Biobehav Rev. 2024 Feb;157:105509. doi: 10.1016/j.neubiorev.2023.105509. Epub 2023 Dec 13. PMID 38101590
- [Result] Chan HH, Hogue O, Mathews ND, Hunter JG, Kundalia R, Hermann JK, Floden DP, Machado AG, Baker KB. Deep cerebellar stimulation enhances cognitive recovery after prefrontal traumatic brain injury in rodent. Exp Neurol. 2022 Sep;355:114136. doi: 10.1016/j.expneurol.2022.114136. Epub 2022 Jun 3. PMID 35667396
- [Result] Olivito G, Serra L, Marra C, Di Domenico C, Caltagirone C, Toniolo S, Cercignani M, Leggio M, Bozzali M. Cerebellar dentate nucleus functional connectivity with cerebral cortex in Alzheimer's disease and memory: a seed-based approach. Neurobiol Aging. 2020 May;89:32-40. doi: 10.1016/j.neurobiolaging.2019.10.026. Epub 2020 Jan 15. PMID 32081466
- [Result] Tacyildiz AE, Bilgin B, Gungor A, Ucer M, Karadag A, Tanriover N. Dentate Nucleus: Connectivity-Based Anatomic Parcellation Based on Superior Cerebellar Peduncle Projections. World Neurosurg. 2021 Aug;152:e408-e428. doi: 10.1016/j.wneu.2021.05.102. Epub 2021 May 29. PMID 34062299
- [Result] Benarroch E. What Is the Role of the Dentate Nucleus in Normal and Abnormal Cerebellar Function? Neurology. 2024 Aug 13;103(3):e209636. doi: 10.1212/WNL.0000000000209636. Epub 2024 Jul 2. No abstract available. PMID 38954796
- [Result] Di Nuzzo C, Ruggiero F, Cortese F, Cova I, Priori A, Ferrucci R. Non-invasive Cerebellar Stimulation in Cerebellar Disorders. CNS Neurol Disord Drug Targets. 2018;17(3):193-198. doi: 10.2174/1871527317666180404113444. PMID 29623859
- [Result] van Dun K, Mitoma H, Manto M. Cerebellar Cortex as a Therapeutic Target for Neurostimulation. Cerebellum. 2018 Dec;17(6):777-787. doi: 10.1007/s12311-018-0976-8. PMID 30276522
- [Result] Manto M, Kakei S, Mitoma H. The critical need to develop tools assessing cerebellar reserve for the delivery and assessment of non-invasive cerebellar stimulation. Cerebellum Ataxias. 2021 Jan 4;8(1):2. doi: 10.1186/s40673-020-00126-w. PMID 33397496
- [Result] Arleo A, Bares M, Bernard JA, Bogoian HR, Bruchhage MMK, Bryant P, Carlson ES, Chan CCH, Chen LK, Chung CP, Dotson VM, Filip P, Guell X, Habas C, Jacobs HIL, Kakei S, Lee TMC, Leggio M, Misiura M, Mitoma H, Olivito G, Ramanoel S, Rezaee Z, Samstag CL, Schmahmann JD, Sekiyama K, Wong CHY, Yamashita M, Manto M. Consensus Paper: Cerebellum and Ageing. Cerebellum. 2024 Apr;23(2):802-832. doi: 10.1007/s12311-023-01577-7. Epub 2023 Jul 10. PMID 37428408
- [Result] Jacobs HIL, Hopkins DA, Mayrhofer HC, Bruner E, van Leeuwen FW, Raaijmakers W, Schmahmann JD. The cerebellum in Alzheimer's disease: evaluating its role in cognitive decline. Brain. 2018 Jan 1;141(1):37-47. doi: 10.1093/brain/awx194. PMID 29053771
- [Result] Liang KJ, Carlson ES. Resistance, vulnerability and resilience: A review of the cognitive cerebellum in aging and neurodegenerative diseases. Neurobiol Learn Mem. 2020 Apr;170:106981. doi: 10.1016/j.nlm.2019.01.004. Epub 2019 Jan 7. PMID 30630042
- [Result] Thal DR, Rub U, Orantes M, Braak H. Phases of A beta-deposition in the human brain and its relevance for the development of AD. Neurology. 2002 Jun 25;58(12):1791-800. doi: 10.1212/wnl.58.12.1791. PMID 12084879
- [Result] Nelson PT, Alafuzoff I, Bigio EH, Bouras C, Braak H, Cairns NJ, Castellani RJ, Crain BJ, Davies P, Del Tredici K, Duyckaerts C, Frosch MP, Haroutunian V, Hof PR, Hulette CM, Hyman BT, Iwatsubo T, Jellinger KA, Jicha GA, Kovari E, Kukull WA, Leverenz JB, Love S, Mackenzie IR, Mann DM, Masliah E, McKee AC, Montine TJ, Morris JC, Schneider JA, Sonnen JA, Thal DR, Trojanowski JQ, Troncoso JC, Wisniewski T, Woltjer RL, Beach TG. Correlation of Alzheimer disease neuropathologic changes with cognitive status: a review of the literature. J Neuropathol Exp Neurol. 2012 May;71(5):362-81. doi: 10.1097/NEN.0b013e31825018f7. PMID 22487856
- [Result] Long JM, Holtzman DM. Alzheimer Disease: An Update on Pathobiology and Treatment Strategies. Cell. 2019 Oct 3;179(2):312-339. doi: 10.1016/j.cell.2019.09.001. Epub 2019 Sep 26. PMID 31564456
- [Result] Sun Z, Zhang X, So KF, Jiang W, Chiu K. Targeting Microglia in Alzheimer's Disease: Pathogenesis and Potential Therapeutic Strategies. Biomolecules. 2024 Jul 11;14(7):833. doi: 10.3390/biom14070833. PMID 39062547
- [Result] Congdon EE, Ji C, Tetlow AM, Jiang Y, Sigurdsson EM. Tau-targeting therapies for Alzheimer disease: current status and future directions. Nat Rev Neurol. 2023 Dec;19(12):715-736. doi: 10.1038/s41582-023-00883-2. Epub 2023 Oct 24. PMID 37875627
- [Result] GBD 2019 Dementia Forecasting Collaborators. Estimation of the global prevalence of dementia in 2019 and forecasted prevalence in 2050: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2022 Feb;7(2):e105-e125. doi: 10.1016/S2468-2667(21)00249-8. Epub 2022 Jan 6. PMID 34998485
- [Result] Scheltens P, De Strooper B, Kivipelto M, Holstege H, Chetelat G, Teunissen CE, Cummings J, van der Flier WM. Alzheimer's disease. Lancet. 2021 Apr 24;397(10284):1577-1590. doi: 10.1016/S0140-6736(20)32205-4. Epub 2021 Mar 2. PMID 33667416